CLINICAL TRIAL: NCT01449578
Title: A Randomized, Blinded, Placebo-Controlled Ascending Dose Study of the Safety and Pharmacokinetics of Dexpramipexole in Healthy Volunteers
Brief Title: Dexpramipexole SAD/MAD Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 223HV103
Record Dates: First submitted 2011-09-22; First posted 2011-10-10 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Dexpramipexole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Part A, Treatment 1 (Experimental): Dexpramipexole single dose (SAD Dose 1)
  Interventions: Drug: Dexpramipexole
- Part A, Treatment 1 placebo (Placebo Comparator): Dexpramipexole single dose placebo (SAD Dose 1)
  Interventions: Drug: Dexpramipexole Placebo
- Part A, Treatment 2 (Experimental): Dexpramipexole single dose (SAD Dose 2)
  Interventions: Drug: Dexpramipexole
- Part A, Treatment 2 placebo (Placebo Comparator): Dexpramipexole single dose placebo (SAD Dose 2)
  Interventions: Drug: Dexpramipexole Placebo
- Part A, Treatment 3 (Experimental): Dexpramipexole single dose (SAD Dose 3)
  Interventions: Drug: Dexpramipexole
- Part A, Treatment 3 placebo (Placebo Comparator): Dexpramipexole single dose placebo (SAD Dose 3)
  Interventions: Drug: Dexpramipexole Placebo
- Part B, Treatment 1 (Experimental): Dexpramipexole multiple dose (MAD Dose 1)
  Interventions: Drug: Dexpramipexole
- Part B, Treatment 1 placebo (Placebo Comparator): Dexpramipexole multiple dose placebo (MAD Dose 1)
  Interventions: Drug: Dexpramipexole Placebo
- Part B, Treatment 2 (Experimental): Dexpramipexole multiple dose (MAD Dose 2)
  Interventions: Drug: Dexpramipexole
- Part B, Treatment 2 placebo (Placebo Comparator): Dexpramipexole multiple dose placebo (MAD Dose 2)
  Interventions: Drug: Dexpramipexole Placebo

INTERVENTIONS:
Drug: Dexpramipexole — Oral Tablet at varying doses
  Other Names: BIIB050
  Arms: Part A, Treatment 1; Part A, Treatment 2; Part A, Treatment 3; Part B, Treatment 1; Part B, Treatment 2
Drug: Dexpramipexole Placebo — Oral tablet at varying doses
  Arms: Part A, Treatment 1 placebo; Part A, Treatment 2 placebo; Part A, Treatment 3 placebo; Part B, Treatment 1 placebo; Part B, Treatment 2 placebo

SUMMARY:
This Phase 1 study will explore the safety, tolerability, and pharmacokinetics of single doses ranging from 300 to 600 mg and multiple daily doses ranging from 225 mg to 300 mg BID dexpramipexole in healthy volunteers.

DETAILED DESCRIPTION:
Preclinical and clinical data to date support the exploration of doses of dexpramipexole higher than 150 mg twice daily for their effectiveness in slowing the progression of ALS. Exploration of doses of dexpramipexole higher than 150 mg twice daily is justified by preclinical and clinical data that suggest that higher doses could potentially be more effective in slowing the progression of ALS than the dose of dexpramipexole currently being explored in Phase 3 studies (150 mg twice daily).

This is a Phase 1, single-center, blinded, randomized, placebo controlled, ascending-dose study consisting of 2 parts; Part A (single-ascending dose [SAD]) and Part B (multiple ascending dose [MAD]). The study will explore safety, tolerability, and pharmacokinetics of single doses ranging from 300 to 600 mg and multiple daily doses ranging from 225 mg to 300 mg BID dexpramipexole in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent.
* Adult males/females aged 18 to 55 years inclusive and between 19 and 30 kg/m2 body mass index (BMI), inclusive at screening.
* Subjects who are healthy as determined by prestudy medical history, physical examination and 12-lead ECG.
* Subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 1 month (females) or 3 months (males) after their last dose of study treatment.
* Normal systemic blood pressure defined as a systolic blood pressure of 90 to 140 mmHg and a diastolic blood pressure of 50 to 90 mmHg.

Exclusion Criteria:

* History of cardiovascular disease (e.g., hypertension, arrhythmia, heart failure, Long QT Syndrome, or other conditions/diseases causing prolongation of the QT/QTc interval).
* A prolongation of QT/QTc interval (e.g., repeated demonstration of a QT/QTc interval >450 ms before study treatment administration) at screening, admission or pre-dose on Day 1.
* Any clinically important abnormalities in resting ECG that may interfere with the interpretation of QTc interval changes at screening, admission or pre-dose on Day 1.
* Prior exposure to dexpramipexole.
* Treatment with pramipexole or any dopamine agonist within 1 year.
* Treatment with another investigational drug or approved therapy for investigational use within 30 days, or 5 half-lives (whichever is longer), or in follow up for any other drug, biologic, or device study.
* Currently active infection or serious infection (e.g., pneumonia, septicemia) within the 2 months prior to Day -2 as determined by the Investigator.
* Female subjects who are pregnant, currently breastfeeding, or attempting to conceive during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability based on medical review of adverse events & results of vital sign measurements, electrocardiogram (ECGs), physical examinations and clinical laboratory tests. | Change from baseline to 11 Days.

SECONDARY OUTCOMES:
Dexpramipexole pharmacokinetics time frame in plasma | pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Overland Park, Kansas, United States